CLINICAL TRIAL: NCT03240692
Title: Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression (SAINT-TRD)
Brief Title: Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression: OL Cohort
Acronym: SAINT-TRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Schatzberg, Alan, M.D. (Individual)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor of Psychiatry & Behavioral Sciences, Director of the Brain Stimulation Laboratory at Stanford University School of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 33797
Record Dates: First submitted 2016-04-23; First posted 2017-08-07 (Actual); Results first posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Treatment Resistant Depression
Keywords: Major Depressive Disorder; Treatment-Resistant Depression; Transcranial Magnetic Stimulation (TMS); Theta-Burst Stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated theta burst treatment (Experimental): All participants will receive theta-burst TMS.
  Interventions: Device: Accelerated theta-burst stimulation treatment

INTERVENTIONS:
Device: Accelerated theta-burst stimulation treatment — All participants will receive intermittent theta-burst stimulation (iTBS) to the left dorsal lateral prefrontal cortex (L-DLPFC). The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered to L-DLPFC using the Magventure Magpro X100 and/or the NextStim TMS system.

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for treatment-resistant depression. In this open label study, all participants will receive accelerated theta-burst stimulation.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is an established technology as therapy for treatment-resistant depression. The approved method for treatment is 10Hz stimulation for 40 minutes over the left dorsolateral prefrontal cortex (L-DLPFC) for a 6 week treatment course. This methodology has been successful for many people with treatment-resistant depression. One of the limitations of this approach is the long duration of the treatment course (approximately a 6 weeks per treatment course). Recently, researchers have aggressively pursued modifying the treatment parameters to reduce treatment course time with some preliminary success. This study intends to further modify the parameters to create a more rapid form of the treatment. This study will also look at the change in neuroimaging biomarkers associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 22 to 80 years of age.
* Able to provide informed consent.
* Diagnosed with Major Depressive Disorder (MDD) and currently experiencing a Major Depressive Episode (MDE).
* Participants may currently be on a stable and adequate dose of an antidepressant therapy but the medication must remain stable throughout study enrollment.
* Participants may also have a history of intolerance to antidepressant medications. These patients with the intolerance history will not be required to be currently taking an antidepressant medication.
* Meet the threshold on the total HAMD17 score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total MADRS score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* Meet the threshold on the total BDI-II score of >/=20 at both screening and baseline visits (Day -5/-14 and Day 0).
* In good general health, as ascertained by medical history.
* If female, a status of non-childbearing potential or use of an acceptable form of birth control.
* Concurrent hypnotic therapy (e.g., with zolpidem, zaleplon, melatonin, or trazodone) will be allowed if the therapy has been stable for at least 4 weeks prior to screening and if it is expected to remain stable.
* History of ECT intolerance is permitted.

Exclusion Criteria:

* Female of childbearing potential who is not willing to use one of the specified forms of birth control during the study.
* Female that is pregnant or breastfeeding.
* Total HAMD score of < 20 at the screen or baseline visits.
* Total MADRS score of < 20 at the screen or baseline visits.
* Total BDI-II score of < 20 at the screen or baseline visits.
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-IV-TR), with the exception of nicotine dependence.
* Current diagnosis of Axis I disorders other than Dysthymic Disorder, Generalized Anxiety Disorder, Social Anxiety Disorder, Panic Disorder, Agoraphobia, or Specific Phobia (unless one of these is comorbid and clinically unstable, and/or the focus of the participant's treatment for the past six months or more).
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes.
* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening.
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation.
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation.
* Positive screening on the urine test for drugs of abuse at screening: cocaine, amphetamines, barbiturates, opiates.
* Current (or chronic) use of opiates.
* History of epilepsy.
* History of shrapnel or metal in the head or skull.
* History of cardiovascular disease or cardiac event.
* History of OCD.
* History of autism spectrum disorder.
* History of rTMS exposure

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Nolan Williams, MD, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
clintrials.gov

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Fox MD, Snyder AZ, Vincent JL, Corbetta M, Van Essen DC, Raichle ME. The human brain is intrinsically organized into dynamic, anticorrelated functional networks. Proc Natl Acad Sci U S A. 2005 Jul 5;102(27):9673-8. doi: 10.1073/pnas.0504136102. Epub 2005 Jun 23. PMID 15976020
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396
- [Derived] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538

RESULTS

PARTICIPANT FLOW:
Groups:
- Accelerated Theta Burst Treatment: All participants will receive theta-burst TMS.
  Accelerated theta-burst stimulation treatment: All participants will receive intermittent theta-burst stimulation (iTBS) to the left dorsal lateral prefrontal cortex (L-DLPFC). The L-DLPFC will be targeted utilizing the Localite neuronavigation system. Stimulation intensity will be standardized at 90% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered to L-DLPFC using the Magventure Magpro X100 and/or the NextStim TMS system.
Period: Overall Study
Arm/Group | Accelerated Theta Burst Treatment
Started | 23
Completed | 21
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.86 (17.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21
Montgomery Asberg Depression Rating Scale (MADRS) Score [Mean (Standard Deviation); unit: Scores on a scale.] — A ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.
  Scores on a scale. | 34.86 (5.29)
Columbia Suicide Severity Rating Scale (C-SSRS) [Mean (Standard Deviation); unit: Scores on a scale.] — A suicidal ideation rating scale created by researchers at Columbia University. The score was calculated by summing the answers to 5 questions. Score range - 0 to 5. Higher score indicate higher suicidal ideation. Population: Participants who provided data are included in the analysis.
  Scores on a scale.
    number analyzed (Participants) | 19
    (all) | 1.42 (0.96)
Hamilton Rating Scale for Depression (HAM-6) [Mean (Standard Deviation); unit: Scores on a scale.] — A 6 item questionnaire used to score the severity of depression. Scale range - 0 to 22 with higher score indicative of greater depressive symptomology.
  Scores on a scale. | 13.90 (2.45)
Hamilton Rating Scale for Depression (HAM-17) [Mean (Standard Deviation); unit: Scores on a scale.] — A provider administered questionnaire used to assess remission and recovery from depression. Scale range - 0 to 52 with higher score indicative of greater depressive symptomology.
  Scores on a scale. | 25.90 (4.79)
Beck Depression Inventory (BDI-II) [Mean (Standard Deviation); unit: Scores on a scale.] — A 21 item Self-report measure of depressive symptoms. Scale range - 0 to 63 with higher score indicative of greater depressive symptomology. Population: Participants who provided data are included in the analysis.
  Scores on a scale.
    number analyzed (Participants) | 18
    (all) | 28.78 (11.68)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Montgomery Asberg Depression Rating Scale (MADRS) Score From Pre-treatment to 1-month
Description: A ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.
Time Frame: Pre-treatment and 1-month post treatment.
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 21
Percentage of change in score | -67.07 (34.71)

2. Secondary Outcome: Percent Change in the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: A suicidal ideation rating scale created by researchers at Columbia University. The score was calculated by summing the answers to 5 questions. Score range - 0 to 5. Higher score indicate higher suicidal ideation.
Time Frame: Pre-treatment to immediately post-treatment (on day 5) and 4 weeks post-treatment
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 19
Percentage of change in score
  Immediately post-treatment: number analyzed (Participants) | 18
  Immediately post-treatment | -100 (0)
  4 weeks post-treatment | -100 (0)

3. Secondary Outcome: Percent Change in the Hamilton Rating Scale for Depression (HAM-6)
Description: A 6 item questionnaire used to score the severity of depression. Scale range - 0 to 22 with higher score indicative of greater depressive symptomology. Additional collection time points were pre-specified; only those time points for which data were collected are reported.
Time Frame: Pre-treatment to immediately post-treatment (on day 5) and 2 weeks,4 weeks and 6 weeks post-treatment
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 21
Percentage of change in score
  immediately post-treatment | -81.96 (25.98)
  Week 2: number analyzed (Participants) | 20
  Week 2 | -71.94 (37.96)
  Week 4: number analyzed (Participants) | 20
  Week 4 | -65.54 (39.40)
  Week 6: number analyzed (Participants) | 1
  Week 6 | -87.5 (0)

4. Secondary Outcome: Percent Change in the Hamilton Rating Scale for Depression (HAM-17)
Description: A provider administered questionnaire used to assess remission and recovery from depression. Scale range - 0 to 52 with higher score indicative of greater depressive symptomology. Additional collection time points were pre-specified; only those time points for which data were collected are reported.
Time Frame: Pre-treatment to immediately post-treatment (on day 5) and 2 weeks, 4 weeks, 6 weeks and 8 weeks post-treatment
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 21
Percentage of change in score
  immediately post-treatment | -81.12 (23.04)
  Week 2: number analyzed (Participants) | 20
  Week 2 | -74.58 (27.97)
  Week 4: number analyzed (Participants) | 20
  Week 4 | -68.25 (32.54)
  Week 6: number analyzed (Participants) | 1
  Week 6 | -88.89 (0)
  Week 8: number analyzed (Participants) | 3
  Week 8 | -93.52 (4.1)

5. Secondary Outcome: Change From Baseline Functional Connectivity to 1-month Post-treatment
Description: We will assess change in resting state fMRI functional connectivity of the subcallosal cingulate to the default mode network and within the default mode network.
Time Frame: Pre-treatment, immediately post-treatment (on day 5), 1-month post-treatment
Population: Data analysis was not possible due to missing data and poor image quality (unable to read)
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Percent Change in the Beck Depression Inventory (BDI-II)
Description: A 21 item Self-report measure of depressive symptoms. Scale range - 0 to 63 with higher score indicative of greater depressive symptomology. Additional collection time points were pre-specified; only those time points for which data were collected are reported.
Time Frame: Pretreatment to immediately post-treatment (on day 5) and 2 weeks, 4 weeks, 6 weeks and 8 weeks post treatment.
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score.
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 18
Percentage of change in score.
  Immediately post-treatment: number analyzed (Participants) | 15
  Immediately post-treatment | -84.89 (15.36)
  Week 2: number analyzed (Participants) | 13
  Week 2 | -65.32 (49.57)
  Week 4: number analyzed (Participants) | 16
  Week 4 | -54.84 (46.85)
  Week 6: number analyzed (Participants) | 2
  Week 6 | -90.74 (13.09)
  Week 8: number analyzed (Participants) | 1
  Week 8 | -100 (0)

7. Secondary Outcome: Percent Change in the Montgomery Asberg Depression Rating Scale (MADRS)
Description: A ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology. Additional collection time points were pre-specified; only those time points for which data were collected are reported.
Time Frame: Pre-treatment to immediately post treatment (on day 5) and 2 weeks, 4 weeks and 8 weeks post-treatment
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of change in score.
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 21
Percentage of change in score.
  immediately post treatment | -85.06 (19.98)
  Week 2 | -78.17 (25.46)
  Week 4: number analyzed (Participants) | 20
  Week 4 | -67.07 (37.74)
  Week 8: number analyzed (Participants) | 2
  Week 8 | -96.30 (5.24)

8. Secondary Outcome: Change From Baseline Functional Connectivity to Immediately Post-treatment
Description: Within subject changes in resting state functional connectivity of subgenual anterior cingulate cortex (sgACC) to default mode network (DMN). frontal (f)DMN (medial prefrontal cortex), median (m)DMN (posterior cingulate cortex and precuneus), left (l)DMN (left angular gyrus), right (r)DMN (right angular gyrus).
  T-statistic (T-score): ratio of departure of estimated value from its hypothesized value to its standard error used in a t-test to determine whether to support or reject the null hypothesis. A T-score of ≥ 2.11 or ≤ -2.11 would be considered a statistically significant change if the accompanying p-value (subject to false discovery rate correction of multiple comparisons) was ≤ 0.05. Positive T-score = increased connectivity, negative T-score = decreased connectivity. No established reference range or clinically meaningful threshold exists for this patient population. Higher connectivity between all DMN nodes to sgACC has been found in depressed vs healthy population.
Time Frame: Pre-treatment to immediately post treatment (on day 5).
Population: Participants who provided data for the respective time point are included in the analysis
Measure: Number; unit: T-score
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 18
T-score
  sgACC-fDMN | -2.335
  sgACC-mDMN | -3.027
  sgACC-lDMN | -2.106
  sgACC-rDMN | -2.660
Statistical Analysis 1: Comparison: Accelerated Theta Burst Treatment; Analysis of subgenual Anterior Cingulate Cortex (sgACC) and frontal Default Mode Network (fDMN) functional connectivity; Test type: Other; p = 0.036, t-test, 2 sided — False Discovery Corrected (FDR) p value. A p-value of ≤ 0.05 was considered to be statistically significant
Statistical Analysis 2: Comparison: Accelerated Theta Burst Treatment; Analysis of subgenual Anterior Cingulate Cortex (sgACC) and medial Default Mode Network (mDMN) functional connectivity; Test type: Other; p = 0.008, t-test, 2 sided — False Discovery Corrected (FDR) p value. A p-value of ≤ 0.05 was considered to be statistically significant
Statistical Analysis 3: Comparison: Accelerated Theta Burst Treatment; Analysis of subgenual Anterior Cingulate Cortex (sgACC) and left Default Mode Network (lDMN) functional connectivity; Test type: Other; p = 0.06, t-test, 2 sided — False Discovery Corrected (FDR) p value. A p-value of ≤ 0.05 was considered to be statistically significant
Statistical Analysis 4: Comparison: Accelerated Theta Burst Treatment; Analysis of subgenual Anterior Cingulate Cortex (sgACC) and right Default Mode Network (rDMN) functional connectivity; Test type: Other; p = 0.017, t-test, 2 sided — False Discovery Corrected (FDR) p value. A p-value of ≤ 0.05 was considered to be statistically significant

9. Other Pre Specified Outcome: A Neuropsychological Test Battery Testing Cognitive Abilities
Description: The Hopkins Verbal Learning Test - Revised (HVLT-DR). Score range 0 to 72, higher score indicates better verbal learning. The Brief Visuospatial Memory Test - Revised (BVMT-DR). Score range 0 to 84, higher score indicates better visuospatial memory. Digit Span test and various tests from the Delis Kaplan Executive Function System (DKEFS) will be used to assess possible cognitive side-effects. Score range 0-36, higher score indicates better executive functions.
Time Frame: Pre-treatment, immediately post-treatment (on day 5) and 4 weeks post-treatment
Population: Participants who provided data for the respective time point are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Accelerated Theta Burst Treatment
Number analyzed (Participants) | 17
score on a scale
  HVLT-DR_Pre-treatment: number analyzed (Participants) | 16
  HVLT-DR_Pre-treatment | 48.81 (6.94)
  HVLT-DR_ immediately post-treatment | 48.18 (9.23)
  HVLT-DR_Week 4: number analyzed (Participants) | 13
  HVLT-DR_Week 4 | 49.77 (10.38)
  BVMT-DR_Pre-treatment | 51.06 (9.44)
  BVMT-DR_ immediately post-treatment | 54.35 (8.14)
  BVMT-DR_Week 4: number analyzed (Participants) | 13
  BVMT-DR_Week 4 | 56.23 (11.02)
  DKEFS_Pre-treatment | 17.35 (4.20)
  DKEFS_ immediately post-treatment | 19.06 (4.13)
  DKEFS_Week 4: number analyzed (Participants) | 13
  DKEFS_Week 4 | 19.15 (3.67)

ADVERSE EVENTS:
Time Frame: Up to 26 weeks.
Arm/Group | Accelerated Theta Burst Treatment
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03240692/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03240692/SAP_002.pdf